CLINICAL TRIAL: NCT01200654
Title: Population Pharmacokinetics of Linezolid in Intensive Care Units Patients Treated for Methicillin-Resistant Staphylococcus Aureus (MRSA) Infections
Brief Title: Population Pharmacokinetics of Linezolid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06 049 02
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Methicillin-Resistant Staphylococcus AureuS
Keywords: Population pharmacokinetics; Linezolid; Monolix; nonlinear mixed effects models
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRSA Infections (Experimental): Methicillin-Resistant Staphylococcus aureus Infections
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — Dosage of 600 mg discontinuous administration twice a day was about studies in safety volunteers
  Other Names: Pharmacokinetics of Linezolid

SUMMARY:
Linezolid is the first of a new class of antibacterial drugs, the oxazolidinones. It has a specific inhibitory activity against Gram positive bacteria, including methicillin-resistant Staphylococcus aureus (MRSA).

Dosage of 600 mg discontinuous administration twice a day was about studies in safety volunteers. The intensive care units patients, with mechanical ventilation, and with severe sepsis, represent highly heterogeneous population responsible of hight variability in pharmacokinetics parameters (augmentation in total volume of distribution, modification in glomerular filtration) wich can lead to antibiotic inefficacy.

In a first time, this study describe the pharmacokinetics of Linezolid in intensive care units patients with severe MRSA infection. The aim of this study is to define and validate a population pharmacokinetic model including the influence of patients' characteristic on the pharmacokinetics of Linezolid.

DETAILED DESCRIPTION:
The demographic, clinical and biological parameters are collected. Patients receive Linezolid as 600 mg twice a day during an administration of 60 minutes.

Blood sampling are collected on the second day after beginning of treatment at the following time : H1, H2, H3, H6 and H12.

The population pharmacokinétics analysis will be carried out using Monolix, a software for the analysis of nonlinear mixed effects models.

ELIGIBILITY:
Inclusion Criteria:

* In-patient stay in intensive care
* Over 18 years old
* Presenting with MRSA nosocomial pneumonia or bacteraemia with a strain thought to be sensitive to Linezolid
* Simplified Acute Physiological Score (SAPS) II > 20
* Expected duration of life > 7 days.

Exclusion Criteria:

* History of allergy to linezolid or any of the antibiotics used
* Isolation of MRSA resistant to linezolid
* Lack of seeds
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The first objective of this study is to research the influence of patients' characteristic on the pharmacokinetics of Linezolid. | Blood sampling are collected on the second day after begining of treatment at the following time : H1, H2, H3, H6 and H12.
  The following demographic, clinical and biological parameters were collected as possible covariates: age, gender, bodyweight, height, etiology of incoming, mechanical ventilation, serum creatinine, proteins, Blood Urea Nitrogen (BUN), leukocyte counts, haemoglobin, C-reactive protein (CRP), and simplified acute physiology scores (SAPS I and II).

SECONDARY OUTCOMES:
The secondary outcome measure are the verification of the clinical and bactériological efficacies, and to look after the residual concentration | At the 48th hours of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Georges, PhMD, Principal Investigator — UH Toulouse